CLINICAL TRIAL: NCT04201106
Title: A Neuroimaging Study of Open-label Placebo in Depressed Adolescents
Acronym: OLP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-29443; R61AT012028 (NIH)
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Depression
Keywords: Placebo; Adolescent Depression; MRI
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): In the control group, the participants will not be taking any placebos or undergoing any other study-related treatments.
- Open Label Placebo Group with Rationale (Experimental)
  Interventions: Behavioral: Open Label Placebo with Rationale
- Open Label Placebo Group without Rationale (Active Comparator)
  Interventions: Behavioral: Open Label Placebo without Rationale

INTERVENTIONS:
Behavioral: Open Label Placebo with Rationale — In the OLP + rationale group, the participants will be prescribed to take placebos for 2 weeks with the standard 4-point accompanying rationale: (1) the placebo effect is powerful, e.g. in clinical trials placebos are roughly 80% as effective as antidepressants; (2) classical conditioning is a possible mechanism for automatic self-healing - meaning that the body can automatically respond to taking placebo pills like Pavlov's dogs who salivated when they heard a bell; (3) placebo-treated patients who are more compliant have better outcomes, therefore the placebos should be taken faithfully; and (4) positive expectations increase placebo effects, but it is OK to have doubts.
  Arms: Open Label Placebo Group with Rationale
Behavioral: Open Label Placebo without Rationale — In the OLP without rationale group, the adolescents will be asked to take placebos for 2 weeks but they will be told that the pills contain inert substance and do not have any pharmacological effect.
  Arms: Open Label Placebo Group without Rationale

SUMMARY:
Major depressive disorder (MDD) is the current leading cause of disability worldwide and adolescence is an especially vulnerable period for the onset of depression. Non-pharmacologic approaches are particularly attractive as treatment of adolescent depression due to the elevated risks of side effects related to the use of psychotropic drugs during development. A recent meta-analysis detected a positive and significant effect of non-deceptive placebos (open-label placebo, OLP) for a series of clinical conditions, including adult depression. To the investigators' knowledge, no studies of OLP have been conducted in depressed adolescents to date, although placebo response rates in adolescent depression are especially high, accounting for over 80% of the actual response to antidepressant treatment. The study's main objective is to estimate the effectiveness and understand the mechanism of OLP in depressed adolescents. The central hypothesis is that the mechanism by which OLP exerts its action in adolescent depression is by forming a positive expectation, which activates endogenous mu-opioid receptor (MOR)-mediated neurotransmission in a network of regions implicated in emotion, stress regulation, and the pathophysiology of MDD, namely, the anterior cingulate cortex (ACC) - striato - amygdalo - thalamic network. The hypothesis has been formulated on the basis of published research and preliminary data. The investigators will test the hypothesis by performing structural and functional neuroimaging in 60 untreated 13-18 year-old adolescents with mild to moderate depression. The proposed research is significant, because it is expected to elucidate the mechanism of action of OLP and advance the understanding of the neural underpinnings of positive expectations in adolescent depression.

DETAILED DESCRIPTION:
This is a randomized controlled study to investigate non-deceptive placebos (open-label placebo, OLP) in depressed adolescents. Participants in this study will be randomly assigned to one of three groups: OLP with the 4-point rationale group (n=20), OLP without rationale group (n=20), and controls (n=20) who will receive the same level of supportive attention from the study clinician. MRI scanning and clinical assessments will be performed at the baseline and after the 2-week treatment or waiting period. The main objective here is to estimate the effectiveness and understand the mechanism of OLP in depressed adolescents. The central hypothesis is that the mechanism by which OLP exerts its action in adolescent depression is by forming a positive expectation, which activates endogenous mu-opioid receptor (MOR)-mediated neurotransmission in a network of regions implicated in emotion, stress regulation, and the pathophysiology of depression, namely, the anterior cingulate cortex (ACC) - striato - amygdalo - thalamic network. The investigators plan to test the central hypothesis in 60 13-18 year-old adolescents with mild to moderate depression by pursuing the following Aims:

AIM 1: To test the effectiveness of OLP in depressed adolescents. Depressed adolescents will be randomly assigned for two weeks to an OLP with the 4-point rationale group (n=20), OLP without rationale group (n=20), and controls (n=20) who will receive the same level of supportive attention from the study clinician. Hypothesis 1: The improvement in depression symptoms measured by the self-report Reynolds Adolescent Depression Scale (RADS-2) in the OLP + rationale group (that combines conscious positive expectation with conditioned response to the ingestion of medication) will be higher than in the OLP without rationale group (conditioned response only) and controls. Positive expectation of recovery will be assessed before and after group assignment and accounted for in the analyses.

AIM 2: To measure neural response to OLP. The OLP groups will receive the first dose of the OLP in the MRI scanner and changes in the cerebral blood perfusion (CBP) will be measured using arterial spin labeling (ASL) MRI. Mechanistically, the investigators expect that the MOR-mediated neurotransmission activated by placebo will be associated with a CBP increase, specifically: Hypothesis 2a: The CBP increase in the ACC - striato - amygdalo - thalamic network after the administration of the OLP + rationale to be higher than in the OLP group and controls. Hypothesis 2b: This CBP increase will correlate with the improvement in RADS-2 scores after two weeks.

AIM 3: To test neural network normalization in depressed adolescents (by comparing to the existing database of MRI scans of healthy teens). The second MRI will be performed after the two weeks. Mechanistically, the investigators expect that through the regular activation by OLP, myelination of the ACC - striato - amygdalo - thalamic network will increase, leading to a normalization of the previously demonstrated hypoconnectivity. Hypothesis 3: The increases in structural and functional connectivity of the ACC - striato - amygdalo - thalamic network after two weeks will correlate with decreases in RADS-2 depression total scores.

ELIGIBILITY:
Inclusion Criteria:

The investigators will include adolescents with mild to moderate depression who meet the following criteria.

* Unmedicated 13-18 year-old adolescents of both sexes with mild to moderate depression, i.e. depressive symptoms corresponding to RADS-2 t-scores of 61-69, under the care of a mental health professional or a primary care doctor.
* Fluency in English

Exclusion Criteria:

* Subjects younger or older than 13-18 years old.
* Psychiatric comorbidities other than anxiety disorder, severe suicidal ideation
* MRI contraindications (ferromagnetic objects on or inside the body, e.g. braces) and pregnancy.
* Potential subjects with an inability or unwillingness to give written informed assent whose legal guardian/representative are unable or unwilling to give written informed consent will be excluded and not allowed to enroll in the study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2032-12-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Reynolds Adolescent Depression Scale (RADS-2) Scores | Baseline and 2 weeks post baseline
  The investigators will be looking at changes in the RADS-2 scores scores. RADS-2 was selected as the primary clinical outcome measure because it is a widely used, well-established, and standardized self-report measure of adolescent depression. The RADS-2 has a possible range of 30 to 120. Higher scores represent higher levels of depression.
The cerebral blood perfusion (CBP) in the anterior cingulate cortex (ACC)- striato - amygdalo - thalamic network | At Baseline
  Blood perfusion in a network of regions implicated in emotion, stress regulation, and the pathophysiology of depression, measured using MRI, specifically, an MRI technique known as arterial spin labeling (ASL).

SECONDARY OUTCOMES:
Change in structural connectivity of the ACC - striato - amygdalo - thalamic network | Baseline and at 2 weeks post baseline
  Brain connectivity in a network of regions implicated in emotion, stress regulation, and the pathophysiology of depression, measured using MRI, specifically, diffusion MRI.
Change in functional connectivity of the ACC - striato - amygdalo - thalamic network | Baseline and at 2 weeks post baseline
  Brain connectivity in a network of regions implicated in emotion, stress regulation, and the pathophysiology of depression, measured using MRI, specifically, functional MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Tony T Yang, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No